CLINICAL TRIAL: NCT05133830
Title: A Two-part, Phase 1, Open-label, Randomized, Parallel-arm, Fixed Sequence, Drug-drug Interaction Study to Investigate the Effect of Linerixibat on Plasma Concentrations of Obeticholic Acid and Conjugates in Healthy Adult Participants
Brief Title: Linerixibat and Obeticholic Acid Drug Interaction Study in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213688
Expanded Access: NCT05448170 (Available)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pruritus
Keywords: Drug-drug interaction; Healthy Volunteers; Linerixibat; Obeticholic acid; Pharmacokinetics
MeSH Terms: conditions — Pruritus | interventions — obeticholic acid

STUDY DESIGN:
Intervention Model Description: Two arms will be evaluated in parallel in Part A. After Part A, if Part B is conducted, one of the two remaining arms will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Arm 1 (Experimental): Participants will receive OCA at dose level 1, 4 hours after the linerixibat administration
  Interventions: Drug: Obeticholic acid; Drug: Linerixibat
- Treatment Arm 2 (Experimental): Participants will receive OCA at dose level 2 along with linerixibat
  Interventions: Drug: Obeticholic acid; Drug: Linerixibat
- Treatment Arm 3 (Experimental): Participants will receive OCA at dose level 1 along with linerixibat
  Interventions: Drug: Obeticholic acid; Drug: Linerixibat
- Treatment Arm 4 (Experimental): Participants will receive OCA at dose level 2, 4 hours after the linerixibat administration
  Interventions: Drug: Obeticholic acid; Drug: Linerixibat

INTERVENTIONS:
Drug: Obeticholic acid — OCA will be administered
Drug: Linerixibat — Linerixibat will be administered

SUMMARY:
This study aims to investigate the effect of linerixibat on plasma concentrations of obeticholic acid (OCA) and its conjugates in healthy adult participants to inform the potential for drug interaction with coadministration of linerixibat and OCA.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or female participants 18 to 50 years of age inclusive, at the time of signing the informed consent
* Body weight greater than (>) 50 kilogram (kg) and body mass index (BMI) within the range 18.5 - 32 kilogram per meter square (kg/m^2) (inclusive)
* Capable of giving signed informed consent as the protocol.

Exclusion Criteria:

* Any active dermatologic disorder leading to or with the potential to cause itching or a recent history of unexplained clinically significant itching locally or generally within the prior 3 months
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) and/or confirmed hepatocellular carcinoma or biliary cancer
* History of gall bladder removal
* Current symptomatic gallstones or inflammatory gall bladder disease
* Significant history of or current disorders that can significantly alter the absorption, metabolism, or elimination of drugs
* Current clinically significant diarrhea
* History of gastrointestinal surgery with ileal resection or ileal bypass at any time
* Any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Administration of any other ileal bile acid transport (IBAT) inhibitor (including linerixibat) or Ocaliva in the 3 months prior to screening
* Past or intended use of over-the-counter or prescription medication, including vitamins and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inhibitor) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless approved by the Investigator in conjunction with GSK
* Current enrolment in a clinical trial or recent participation in a clinical trial and has received an investigational product within 30 days before the first dose in the current study
* Exposure to more than 4 new chemical entities within 12 months before the first dose in the current study
* Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5x upper limit of normal (ULN)
* Bilirubin >1.5xULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin lesser than (<)35%
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test or positive hepatitis C riboneucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention
* Positive pregnancy test at screening or at Day -1
* Positive human immunodeficiency virus (HIV) antibody test
* QT interval corrected (QTc) >450 millisecond (msec)
* Regular use of known drugs of abuse or history of drug abuse or dependence within 6 months of the study
* Participants with moderate (or greater) alcohol consumption
* History of or regular use of tobacco- or nicotine-containing products in the 3 months prior to screening.
* Female participants unable or unwilling to comply with specific contraception restrictions as detailed in the protocol
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within a 56-day period
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Average trough concentration (Ctrough) in plasma for total-OCA at steady state | Days 35 to 38

SECONDARY OUTCOMES:
Area under the concentration curve from time 0 to t (AUC0-t) for OCA, tauro-OCA, glyco-OCA and total-OCA at steady state | At Day 18 and Day 37
AUC from time 0 to 24 hour (AUC0-24) for OCA, tauro-OCA, glyco-OCA and total-OCA at steady state | Up to 24 hours on Day 18 and Day 37
Maximum observed plasma concentration (Cmax) for OCA, tauro-OCA, glyco-OCA and total-OCA at steady state | At Day 18 and Day 37
Average trough concentration (Ctrough) in plasma for OCA, tauro-OCA, glyco-OCA and total-OCA at steady state | Days 17 to 19 and Days 35 to 38
Time to maximum concentration (Tmax) for OCA, tauro-OCA, glyco-OCA and total-OCA | At Day 18 and Day 37
Ctrough of total OCA over Days 17 to 19 and Days 35 to 38 | Days 17 to 19 and Days 35 to 38
Number of participants with adverse events | Up to Day 52

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com